CLINICAL TRIAL: NCT05319392
Title: Exploring the Transcriptomic Signatures and Their Relevance in Gastric Adenocarcinoma
Brief Title: Transcriptomic Signatures in Gastric Adenocarcinoma
Acronym: GAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, raghavendra, Assistant professor (Clinical chemistry), Sanjay Gandhi Postgraduate Institute of Medical Sciences
Other Study IDs: 2021-240-PhD-EXP-42
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Gastric Adenocarcinoma
Keywords: Gastric cancer; Tumor microenvironment; Transcriptomics; Differential gene expression
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Surgically resected fresh tissue samples and FFPE blocks of surgical specimens from gastric adenocarcinoma patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Gastric Adenocarcinoma: Patients with origin of tumor in distal part of stomach who underwent total or partial gastrectomy after biopsy examination with availability of follow-up and archived FFPE tissue will be considered for this study.
  Interventions: Diagnostic Test: Observational study

INTERVENTIONS:
Diagnostic Test: Observational study — Exploration of transcriptomic signatures related to tumor microenvironment having a significant role in prognosis of gastric adenocarcinoma patients

SUMMARY:
Gastric Adenocarcinoma (GAC) accounting for the major percentage of all stomach malignancies is associated with a poor overall survival of 25-30% despite the advancement in treatment strategies. Several factors associated with tumor microenvironment (TME) are thought to play an important role in tumorigenesis and acquired chemoresistance to therapies that are not otherwise addressed by the comprehensive molecular classification of GAC given by TCGA and ACRG. In the present study investigators intend to do transcriptome profiling of GAC tumor tissue and adjacent normal tissue to investigate differentially expressed genes between the two in relation to TME which might help in identification of gene signatures that are clinically relevant with survival outcome in Gastric Adenocarcinoma.

DETAILED DESCRIPTION:
This study on Gastric adenocarcinoma is retrospective as well as prospective that will be conducted at SGPGIMS, Lucknow, India. Patients undergoing gastric resection at the department of surgical gastroenterology who are diagnosed with GAC based on the endoscopic biopsy in the department of pathology will be recruited for the study. For the retrospective part of study, cases will be selected based on histological findings retrieved from hospital information system and patient records.

For sample collection, surgically resected fresh specimens will be collected in RNAlater and stored at -80⁰C. Archived formalin fixed paraffin embedded (FFPE) tissue blocks for retrospective cases will be retrieved and reviewed histopathologically. After a confirmed diagnosis of GAC, tissues will be processed to obtain tumor and normal tissue for experimental part.

RNA from the tumor and normal area will be extracted from FFPE blocks and fresh tissue specimens. Whole transcriptomic next generation sequencing will be performed after successful quality check, library preparation and amplification. The gene expression data obtained from sequencing will be bioinformatically analyzed to elucidate differential gene expression between tumor and adjacent normal tissue in relation to TME. The significantly differentially expressed genes between the tumor and normal areas will be annotated and identified using bioinformatic packages for gene annotation. Using statistical analysis, the differentially expressed genes will be correlated with the patient's clinical features and outcome to identify TME genes with significant prognostic value.

ELIGIBILITY:
Inclusion Criteria:

* Patients with origin of tumor in distal part of stomach
* Patients who underwent Total or partial Gastrectomy after Biopsy examination
* Availability of follow up in Radiotherapy or Gastro department
* Availability of FFPE gastrectomy specimen tissue of selected cases in Histopathology

Exclusion Criteria:

* Patients with origin of tumor in proximal part of stomach
* Patients with only biopsy available
* Patients whose follow-up is not available
* Unavailability of FFPE tissue blocks

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with distal Gastric Adenocarcinoma at SGPGIMS will be recruited for this study
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2025-04-06 (Estimated); Study Completion 2025-10-06 (Estimated)

PRIMARY OUTCOMES:
Transcriptome profiling of Gastric adenocarcinoma | Range of 6 months to 5 years of patient recruitment
  To obtain gene expression data of cancerous and normal tissue through RNA - sequencing
Differential gene expression analysis in Gastric adenocarcinoma | Range of 6 months to 5 years of patient recruitment
  To determine differentially expressed gene between tumor and normal tissue through bioinformatic analysis of gene expression data
Influence of tumor microenvironment on gene expression profile of gastric adenocarcinoma | Range of 6 months to 5 years of patient recruitment
  To identify tumor microenvironment related genes and their functional annotation using bioinformatic packages
Correlation of tumor microenvironment related genes with patient's clinical features | Range of 6 months to 5 years of patient recruitment
  To correlate differentially expressed tumor microenvironment related gene with outcome in patients to identify genes significantly related with overall survival

SECONDARY OUTCOMES:
Patient risk stratification based on correlation between gene expression and overall survival | Range of 6 months to 5 years of patient recruitment
  To stratify patients based on gene signatures related to overall survival in gastric adenocarcinoma patients

CONTACTS AND LOCATIONS:
Overall Officials: Raghavendra Lingaiah, Principal Investigator — SGPGIMS
Locations (1):
- Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahn B, Chae YS, Kim CH, Lee Y, Lee JH, Kim JY. Tumor microenvironmental factors have prognostic significances in advanced gastric cancer. APMIS. 2018 Oct;126(10):814-821. doi: 10.1111/apm.12889. PMID 30264431
- [Background] Zhang S, Zeng Z, Liu Y, Huang J, Long J, Wang Y, Peng X, Hu Z, Ouyang Y. Prognostic landscape of tumor-infiltrating immune cells and immune-related genes in the tumor microenvironment of gastric cancer. Aging (Albany NY). 2020 Sep 23;12(18):17958-17975. doi: 10.18632/aging.103519. Epub 2020 Sep 23. PMID 32969836
- [Background] Qiu XT, Song YC, Liu J, Wang ZM, Niu X, He J. Identification of an immune-related gene-based signature to predict prognosis of patients with gastric cancer. World J Gastrointest Oncol. 2020 Aug 15;12(8):857-876. doi: 10.4251/wjgo.v12.i8.857. PMID 32879664
- [Background] Ren N, Liang B, Li Y. Identification of prognosis-related genes in the tumor microenvironment of stomach adenocarcinoma by TCGA and GEO datasets. Biosci Rep. 2020 Oct 30;40(10):BSR20200980. doi: 10.1042/BSR20200980. PMID 33015704
- [Background] Cai WY, Dong ZN, Fu XT, Lin LY, Wang L, Ye GD, Luo QC, Chen YC. Identification of a Tumor Microenvironment-relevant Gene set-based Prognostic Signature and Related Therapy Targets in Gastric Cancer. Theranostics. 2020 Jul 9;10(19):8633-8647. doi: 10.7150/thno.47938. eCollection 2020. PMID 32754268
- [Background] Li T, Gao X, Han L, Yu J, Li H. Identification of hub genes with prognostic values in gastric cancer by bioinformatics analysis. World J Surg Oncol. 2018 Jun 19;16(1):114. doi: 10.1186/s12957-018-1409-3. PMID 29921304